CLINICAL TRIAL: NCT04565951
Title: Increasing Help-Seeking Behavior Among Transitioning Veterans at Risk for Suicide With Online Gatekeeper Training: A Pilot Study of PsychArmor S.A.V.E.
Brief Title: Increasing Help-Seeking Behavior Among Transitioning Veterans at Risk for Suicide With Online Gatekeeper Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Canandaigua VA Medical Center (U.S. Federal Agency); PsychArmor Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PPO 20-166; HX003249 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2020-09-21; First posted 2020-09-28 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-09

CONDITIONS: Suicide Prevention
Keywords: suicide; suicide prevention; mental health; veterans
MeSH Terms: conditions — Suicide Prevention; Suicide; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either the intervention or the control group. Block-randomization schemes using random block sizes to assign the two study arms will be created in R using the blockrand package before study start and pre-loaded into survey software. The intervention, called VA S.A.V.E., is an online, video-based training tailored to veterans and their close supports. The control group will consist of a "sham" training - a different online, video-based training course developed by the PsychArmor Institute for military service members, veterans, and their loved ones. Topics in this "sham" training may include information relevant to transitioning veterans and their loved ones, such as preparing finances, networking, searching for a job, and using educational benefits. The length of the training will be matched to the intervention (24 minutes) and the "sham" training will also contain other design features similar to the intervention (e.g., motion graphics).
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded by limiting details about the study hypotheses and differences between the study arms. Blinding will also be achieved because no study personnel are involved in intervention delivery. The biostatistician will be blinded for analyses involving study group comparisons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Participants in this arm will receive the intervention, VA S.A.V.E.
  Interventions: Behavioral: VA S.A.V.E.
- Sham arm (Sham Comparator): Participants in this arm will receive a "sham" training, not the intervention, consisting of information unrelated to suicide prevention but relevant to transitioning veterans and their loved ones.
  Interventions: Behavioral: Sham intervention

INTERVENTIONS:
Behavioral: VA S.A.V.E. — The intervention is called VA S.A.V.E. It is an online video-based training tailored to veterans and their close supports. It is free, brief (24 minutes), and includes three scripted role plays.
  Arms: Treatment arm
Behavioral: Sham intervention — A "sham" training consisting of information unrelated to suicide prevention but relevant to transitioning veterans and their loved ones.
  Arms: Sham arm

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of a gatekeeper training called VA S.A.V.E. which was developed through a partnership between the VA and the PsychArmor Training Institute. Gatekeeper training teaches "gatekeepers" skills in how to identify a person with suicide risk, inquire about suicidal thoughts, and help make a connection to professional treatment. VA S.A.V.E. is a brief, novel online gatekeeper training that was created and designed specifically for Veterans and their family and friends. In this study, the investigators will recruit Veterans who have recently transitioned out of the military, as well as their family and friends. Participants in the study will be asked to complete a survey, watch the VA S.A.V.E. training, and complete several follow-up surveys over six months. A small subset of participants will also be invited to participate in an interview.

DETAILED DESCRIPTION:
Background: Suicide is an urgent public health crisis, and transitioning Veterans (those who have recently separated from the military) are a high-risk group for suicide. A key component to advancing suicide prevention efforts among at-risk Veterans is to address low levels of help-seeking and engagement in treatment, including Veterans Health Administration (VHA) care. Veterans are most likely to disclose suicidal thoughts to their close supports-family members, friends, and their peers. However, Veterans and their close supports rarely receive training in how to help a peer at risk of suicide, despite strong interest in such training. Gatekeeper training is a key strategy with potential to help address these challenges. Gatekeeper training teaches "gatekeepers" skills in how to identify a Veteran with suicide risk, inquire about suicidal thoughts, and help make a connection to professional treatment; it may benefit the trainee's own mental health too. VA S.A.V.E., developed through a partnership between the VA and the PsychArmor Training Institute, is a brief, novel online gatekeeper training designed for Veterans and their close supports.

Significance/Impact: This project focuses on VA's topic clinical priority, suicide prevention. The 2019 VA and Department of Defense Clinical Practice Guidelines also identified gatekeeper training as an important research gap and priority for future research. This research design addresses three separate goals and objectives contained in VA's National Strategy for Preventing Veteran Suicide, including involvement of Veterans' close supports.

Innovation: This proposal employs the novel approach of recruiting Veterans and their close supports through online social media advertisements, allowing for broad outreach, suicide prevention targeting Veterans outside the VA network, and the potential to test the effectiveness of gatekeeper training on a large scale. Online gatekeeper trainings are highly scalable public health strategies with the potential to diffuse through online social networks.

Specific Aims: The primary objective is to conduct a pilot randomized controlled trial (RCT) to evaluate the feasibility and acceptability of the online gatekeeper training VA S.A.V.E. To reach this objective the investigators will achieve these aims: 1) Determine the feasibility of recruiting participants via social media, engaging them to participate in an online gatekeeper training program, and retaining them in an online intervention study; and 2) Determine the acceptability of VA S.A.V.E. in a pilot RCT, and evaluate measures for use in a future larger-scale RCT.

Methodology: This is a two-arm pilot randomized clinical trial involving 200 participants. Participants will be recruited through social media advertisements targeting transitioning Veterans and their close supports (family and friends). Participants will be randomized to take the VA S.A.V.E. gatekeeper training or a "sham" control training and followed for 6 months. Mixed quantitative and qualitative methods will be used to assess outcomes on feasibility and acceptability. Additional data collection and analysis of measures related to suicide prevention, such as gatekeeper behaviors, knowledge, stigma, self-efficacy, and social norms measures will help prepare for a larger-scale RCT.

Implementation/Next Steps: By using an extremely scalable intervention and building off existing VA practices and partnerships, this project will be very well-positioned for further evaluation and implementation into VA practice if found to be effective. It is freely available online, making it highly amenable to being rapidly taken to scale. Results of this project will inform future efforts to disseminate and/or revise VA S.A.V.E.

ELIGIBILITY:
Inclusion Criteria:

* A veteran who has served on active duty in the U.S. Armed Forces within the prior 12 months, OR a person who feels "close to" a veteran; AND
* Social contact with a veteran at least weekly

Exclusion Criteria:

* Lack a U.S. phone number, email, or computer access; OR
* Not fluent in English; OR
* Have previously taken or intend to take VA S.A.V.E. training; OR
* Duplicate study entry or misrepresentation of veteran status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan R. Teo, MD MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teo AR, Call AA, Hooker ER, Fong C, Karras E, Dobscha SK. Feasibility of recruitment and retention in a remote trial of gatekeeper training for close supports of military veterans: Mixed methods study. Contemp Clin Trials Commun. 2022 Sep 5;30:100993. doi: 10.1016/j.conctc.2022.100993. eCollection 2022 Dec. PMID 36159001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via a social media campaign that ran a series of sponsored ads on Facebook from March 13, 2021 to May 24, 2021.
Period: Overall Study
Arm/Group | Sham Arm | Treatment Arm
Started | 151 | 130
Responded to Baseline Survey | 112 | 102
Completed (Responded to 6-month follow-up survey) | 71 | 84
Not Completed | 80 | 46
Not completed — Lost to Follow-up | 66 | 38
Not completed — Withdrawal by Subject | 14 | 7
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 281 participants who enrolled, 214 completed the baseline survey. This group of 214 participants (n=102 in the VA S.A.V.E. arm, and n=112 in the control arm) constituted the primary analytic sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Arm | Treatment Arm | Total
Number analyzed (Participants) | 112 | 102 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (13.8) | 55.6 (12.7) | 54.3 (13.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male/man | 11 | 11 | 22
  Female/woman | 99 | 90 | 189
  Genderqueer/non-binary | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 107 | 97 | 204
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 102 | 90 | 192
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 2 | 4 | 6
Veteran status [Count of Participants; unit: Participants]
  No, never served | 77 | 69 | 146
  Yes, now on active duty | 5 | 3 | 8
  Yes, active duty in the past | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: Number enrolled; proportion of eligible who enroll
Time Frame: baseline (T=0)
Population: For the purposes of assessing the proportion of eligible participants who enroll, this group includes all those who completed the online screener and screened in as eligible.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: This group includes all participants prior to randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 1278
Participants
  Enrolled | 281
  Not enrolled | 997

2. Primary Outcome: Survey Completion Rates
Description: Survey completion at each survey timepoint
Time Frame: 1-month follow-up, 2-month follow-up, 3-month follow-up, 4-month follow-up, 5-month follow-up, 6-month follow-up
Population: This includes all those who completed baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Arm | Treatment Arm
Number analyzed (Participants) | 112 | 102
Participants
  Completed 1-month follow up | 71 | 79
  Completed 2-month follow up | 68 | 82
  Completed 3-month follow up | 63 | 80
  Completed 4-month follow up | 67 | 82
  Completed 5-month follow up | 66 | 78
  Completed 6-month follow up | 71 | 84

3. Secondary Outcome: Training Completion
Description: Percentage of training completed
Time Frame: Post-training (immediately after), approximately 1 hour
Population: All those who at least started the training video are included here.
Measure: Mean (95% Confidence Interval); unit: percentage of video watched
Arm/Group | Sham Arm | Treatment Arm
Number analyzed (Participants) | 112 | 102
percentage of video watched | 66.1 [58.2 to 73.9] | 76.6 [69.3 to 83.8]

4. Secondary Outcome: Satisfaction With the Intervention Video
Description: An 8-item satisfaction questionnaire, adapted from the CSQ-8, where higher scores indicate greater satisfaction. Total scores range from 8 - 32, with higher scores indicating greater satisfaction.
Time Frame: Post-training (immediately after), approximately 1 hour
Population: This includes all those who completed the post-training survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 100
units on a scale | 26.6 (4.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sham Arm | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/151 | 1/130
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/130
Other Adverse Events (participants affected / at risk) | 0/151 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT04565951/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT04565951/ICF_000.pdf